CLINICAL TRIAL: NCT01144416
Title: A Phase 3, Randomized, Double-blind, Active-controlled, Non-inferiority Trial to Investigate the Efficacy and Safety of a Single Injection of SCH 900962 (Corifollitropin Alfa) to Induce Multifollicular Development for Controlled Ovarian Stimulation (COS) Using Daily Recombinant FSH (recFSH) as a Reference in Women Aged 35 to 42 Years (Phase 3; Protocol No. P06029)
Brief Title: Efficacy and Safety Study of a Single Injection of SCH 900962 Versus Daily recFSH Injections in Women Undergoing Controlled Ovarian Stimulation (Study P06029)
Acronym: PURSUE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P06029
Record Dates: First submitted 2010-06-11; First posted 2010-06-15 (Estimated); Results first posted 2012-12-27 (Estimated); Last update posted 2022-02-03 (Actual); Status verified 2022-02

CONDITIONS: Infertility
Keywords: Reproductive Techniques, Assisted; Follicle Stimulating Hormone, Human; Fertilization In Vitro
MeSH Terms: conditions — Infertility; Helping Behavior | interventions — follicle stimulating hormone, human, with HCG C-terminal peptide; follitropin beta

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single injection of 150 µg SCH 900962 (MK-8962) (Experimental): Participants received a single injection of 150 ug SCH 900962 (MK-8962) on Stimulation Day 1 and 7 injections with placebo-recFSH from Stimulation Days 1-7
  Interventions: Biological: SCH 900962 / Corifollitropin alfa / Org 36286; Drug: Placebo for recFSH
- Daily 300 IU recFSH (Active Comparator): Participants received a single injection of placebo SCH 900962 (MK-8962) on Stimulation Day 1 and 7 injections of recFSH from Stimulation Days 1-7
  Interventions: Biological: RecFSH / follitropin beta; Drug: Placebo for SCH 900962

INTERVENTIONS:
Biological: SCH 900962 / Corifollitropin alfa / Org 36286 — SCH 900962 will be provided as ready-for-use prefilled syringes containing 150 μg corifollitropin alfa per 0.5 mL. On day 2 or 3 of the menstrual cycle, a single dose of 150 μg corifollitropin alfa will be administered by subcutaneous injection in the abdominal wall in the morning.
  Other Names: MK-8962
  Arms: Single injection of 150 µg SCH 900962 (MK-8962)
Biological: RecFSH / follitropin beta — RecFSH will be provided as a ready-for-use solution in 900 IU cartridges for subcutaneous injection with the Follistim Pen. Starting on day 2 or 3 of the menstrual cycle (=Stimulation Day 1), administration of recFSH will be done in the morning by daily injections in the abdominal wall. A starting dose of 300 IU will be administered and fixed for at least 7 days.
  Other Names: Follistim® AQ Cartridge
  Arms: Daily 300 IU recFSH
Drug: Placebo for SCH 900962 — Supplied as a pre-filled syringe containing an identical solution when
  compared to SCH 900962, however without the active ingredient corifollitropin alfa. On Day 2 or 3 of the menstrual cycle (=Stimulation Day 1), a single dose of placebo SCH 900962 is to be administered in the morning by subcutaneous injection in the abdominal wall.
  Arms: Daily 300 IU recFSH
Drug: Placebo for recFSH — Supplied as identical ready-for-use solution, but without the active ingredient, in cartridges for subcutaneous injection with the Follistim Pen. Starting on day 2 or 3 of the menstrual cycle (=Stimulation Day 1), administration of placebo-recFSH will be done by daily injections in the abdominal wall in the morning for a period of 7 days.
  Arms: Single injection of 150 µg SCH 900962 (MK-8962)

SUMMARY:
The purpose of this study is to show that a single injection of SCH 900962/MK-8962 is non-inferior to daily injections of recombinant follicle-stimulating hormone (recFSH) during the first week of ovarian stimulation in terms of the number of vital pregnancies (ie, presence of at least one fetus with heart activity as assessed by ultrasound at least 35 days after embryo transfer) in women aged 35 to 42 years undergoing controlled ovarian stimulation (COS) prior to in vitro fertilization (IVF) or intracytoplasmic sperm injection (ICSI).

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent for trial P06029 as well as for the Frozen-Thawed Embryo Transfer (FTET) follow-up trial P06031, and for the pharmacogenetic analysis (if applicable).
* Female and >=35 to <=42 years of age with indication for COS and IVF/ICSI.
* Body weight ≥50.0 kg, body mass index (BMI) >=18.0 to <=32.0 kg/m2.
* Regular spontaneous menstrual cycle with variation not outside the 24-35 days.
* Ejaculatory sperm must be available (donated and/or cryopreserved sperm is allowed).
* Results of clinical laboratory tests, cervical smear, physical examination within normal limits or clinically acceptable to the investigator.
* Adhere to trial schedule.

Exclusion Criteria:

* A recent history of/or any current endocrine abnormality.
* A history of ovarian hyper-response or ovarian hyperstimulation syndrome (OHSS).
* A history of/or current polycystic ovary syndrome.
* More than 20 basal antral follicles <11 mm (both ovaries combined) in the early follicular phase.
* Less than 2 ovaries or any other ovarian abnormality.
* Unilateral or bilateral hydrosalpinx.
* Intrauterine fibroids ≥5 cm or any clinically relevant pathology, which could impair embryo implantation or pregnancy continuation.
* More than three unsuccessful COS cycles for IVF/ICSI since the last established ongoing pregnancy (if applicable).
* A history of non- or low ovarian response to FSH/human menopausal gonadotropin (hMG) treatment.
* A history of recurrent miscarriage.
* FSH >15.0 IU/L or luteinizing hormone (LH) >12.0 IU/L during the early follicular phase.
* Positive for human immunodeficiency virus (HIV) or Hepatitis B.
* Contraindications for the use of gonadotropins or gonadotropin releasing hormone (GnRH) antagonists.
* A recent history of/or current epilepsy, thrombophilia, diabetes, cardiovascular, gastro-intestinal, hepatic, renal or pulmonary or auto-immune disease requiring regular treatment.
* Smoking or recently stopped smoking (ie, within the last 3 months prior to signing informed consent).
* A recent history or presence of alcohol or drug abuse.
* The participant or the sperm donor has known gene defects, genetic abnormalities, or abnormal karyotyping, relevant for the current indication or for the health of the offspring.
* Prior or concomitant medications disallowed by protocol.

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1424 (Actual)
Dates: Start 2010-06; Primary Completion 2011-07 (Actual); Study Completion 2012-04 (Actual)

REFERENCES:
- [Result] Boostanfar R, Shapiro B, Levy M, Rosenwaks Z, Witjes H, Stegmann BJ, Elbers J, Gordon K, Mannaerts B; Pursue investigators. Large, comparative, randomized double-blind trial confirming noninferiority of pregnancy rates for corifollitropin alfa compared with recombinant follicle-stimulating hormone in a gonadotropin-releasing hormone antagonist controlled ovarian stimulation protocol in older patients undergoing in vitro fertilization. Fertil Steril. 2015 Jul;104(1):94-103.e1. doi: 10.1016/j.fertnstert.2015.04.018. Epub 2015 May 21. PMID 26003273
- [Derived] Lawrenz B, Beligotti F, Engelmann N, Gates D, Fatemi HM. Impact of gonadotropin type on progesterone elevation during ovarian stimulation in GnRH antagonist cycles. Hum Reprod. 2016 Nov;31(11):2554-2560. doi: 10.1093/humrep/dew213. Epub 2016 Sep 12. PMID 27619773
- [Derived] Zandvliet AS, Prohn M, de Greef R, van Aarle F, McCrary Sisk C, Stegmann BJ. Impact of patient characteristics on the pharmacokinetics of corifollitropin alfa during controlled ovarian stimulation. Br J Clin Pharmacol. 2016 Jul;82(1):74-82. doi: 10.1111/bcp.12939. Epub 2016 May 31. PMID 26991902
- [Derived] Oehninger S, Nelson SM, Verweij P, Stegmann BJ. Predictive factors for ovarian response in a corifollitropin alfa/GnRH antagonist protocol for controlled ovarian stimulation in IVF/ICSI cycles. Reprod Biol Endocrinol. 2015 Oct 31;13:117. doi: 10.1186/s12958-015-0113-1. PMID 26520396

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women, aged between 35 and 42 years, with an indication for controlled ovarian stimulation and in vitro fertilization/intracytoplasmic sperm injection without a history of previous hyper or low ovarian response to follicle-stimulating hormone/human menopausal gonadotropins, ovarian hyperstimulation syndrome (OHSS), or polycystic ovary syndrome.
Pre-assignment Details: 1424 participants were originally enrolled in the study. All data for 1 participant, who was incorrectly randomized and did not receive study medication and for all 33 participants at 1 clinical site were excluded from all analyses, including disposition, prior to unblinding. Only women who became pregnant continued into Pregnancy Follow-up period.
Groups:
- Single Injection of 150 µg SCH 900962/MK-8962: Participants received a single injection of 150 ug SCH 900962 (MK-8962) on Stimulation Day 1 and 7 injections with placebo-recombinant follicle-stimulating hormone (recFSH) from Stimulation Days 1-7
- Daily 300 IU recFSH: Participants received a single injection of placebo SCH 900962 (MK-8962) on Stimulation Day 1 and 7 injections of 300 IU recFSH from Stimulation Days 1-7
Period: Intervention Period
Arm/Group | Single Injection of 150 µg SCH 900962/MK-8962 | Daily 300 IU recFSH
Started | 694 | 696
Completed | 632 | 647
Not Completed | 62 | 49
Not completed — Adverse Event | 5 | 6
Not completed — Insufficient ovarian response | 11 | 17
Not completed — Risk of OHSS | 0 | 1
Not completed — Too high ovarian response | 4 | 2
Not completed — No/too few/bad oocytes | 7 | 5
Not completed — No or abnormal fertilization | 25 | 10
Not completed — No/too few/bad quality embryos | 3 | 3
Not completed — Other | 7 | 5
Period: Pregnancy Follow-up Period
Arm/Group | Single Injection of 150 µg SCH 900962/MK-8962 | Daily 300 IU recFSH
Started | 154 (Participants received 150 ug SCH 900962 in Intervention Period and became pregnant.) | 167 (Participants received daily injections of 300 IU recFSH in Intervention Period and became pregnant.)
Completed | 146 | 157
Not Completed | 8 | 10

BASELINE CHARACTERISTICS:
Groups:
- Single Injection of 150 µg SCH 900962/MK-8962: Participants received a single injection of 150 ug SCH 900962 (MK-8962) on Stimulation Day 1 and 7 injections with placebo-recFSH from Stimulation Days 1-7
- Total: Total of all reporting groups
Arm/Group | Single Injection of 150 µg SCH 900962/MK-8962 | Daily 300 IU recFSH | Total
Number analyzed (Participants) | 694 | 696 | 1390
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.0 (2.2) | 38.0 (2.2) | 38.0 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 694 | 696 | 1390
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Vital Pregnancy
Description: Vital pregnancy was defined as the presence of at least 1 fetus with heart activity at least 35 days (≥5 weeks) after embryo transfer in the controlled ovarian stimulation (COS) treatment cycle
Time Frame: Vital pregnancy will be assessed by ultrasound at least 35 days after embryo transfer (with a timeframe of 35-42 days). Time from start of study treatment to embryo transfer is maximally 24 days.
Population: Intent-To-Treat Group: all randomized participants who received 1 or more dose(s) of SCH 900962 or recFSH. Participants were grouped according to the treatment they were randomized to. Participants who did not have embryo transfer or who were lost to follow-up before the ultrasound assessment to confirm vital pregnancy were counted as non-pregnant.
Measure: Number; unit: percentage of participants
Arm/Group | Single Injection of 150 µg SCH 900962/MK-8962 | Daily 300 IU recFSH
Number analyzed (Participants) | 694 | 696
percentage of participants | 23.9 | 26.9
Statistical Analysis 1: Comparison: Single Injection of 150 µg SCH 900962/MK-8962 vs Daily 300 IU recFSH; Test type: Non-Inferiority or Equivalence — The pre-defined non-inferiority margin was -8%; generalized linear model; The estimated difference in percentage vital pregnancy was adjusted for age class as stratified (≤38 yrs vs. >38 yrs); Difference in percentage vital pregnancy = -3.0, 95% CI 2-sided [-7.4 to 1.4]

2. Secondary Outcome: Number of Oocytes Retrieved Per Attempt
Description: The number of cumulus oocyte-complexes retrieved was summarized per treatment group and per attempt (= per started COS cycle).
Time Frame: Maximally 21 days after the start of study treatment.
Population: Intent-To-Treat (ITT) Group, defined as all randomized participants who received one or more dose(s) of SCH 900962 or recFSH. Participants were grouped according to the treatment they were randomized to. The number of oocytes retrieved were set to zero for participants who did not have oocyte retrieval.
Measure: Mean (Standard Deviation); unit: Number of oocytes
Arm/Group | Single Injection of 150 µg SCH 900962/MK-8962 | Daily 300 IU recFSH
Number analyzed (Participants) | 694 | 696
Number of oocytes | 10.7 (7.2) | 10.3 (6.8)
Statistical Analysis 1: Comparison: Single Injection of 150 µg SCH 900962/MK-8962 vs Daily 300 IU recFSH; Test type: Non-Inferiority or Equivalence — The pre-defined non-inferiority margin was -3 oocytes; ANOVA; The estimated difference in number of oocytes retrieved was adjusted for age class as stratified (≤38 yrs vs. >38 yrs) and center; Mean Difference (Final Values) = 0.5, 95% CI 2-sided [-0.2 to 1.2]

3. Secondary Outcome: Live Birth Rate
Description: The live-birth rate is the percentage of participants with at least 1 live born infant after an ongoing pregnancy in the controlled ovarian stimulation (COS)treatment cycle relative to the number of participants treated.
Time Frame: Approximately nine months after embryo transfer
Population: Intent-To-Treat Group: all randomized participants who received 1 or more dose(s) of SCH 900962 or recFSH. Participants were grouped according to the treatment they were randomized to.
Measure: Number; unit: Percentage of participants
Arm/Group | Single Injection of 150 µg SCH 900962/MK-8962 | Daily 300 IU recFSH
Number analyzed (Participants) | 694 | 696
Percentage of participants | 21.3 | 23.4
Statistical Analysis 1: Comparison: Single Injection of 150 µg SCH 900962/MK-8962 vs Daily 300 IU recFSH; Test type: Non-Inferiority or Equivalence — The pre-defined non-inferiority margin was -8%; generalized linear model; The estimated difference in live birth rate was adjusted for age class as stratified (≤38 yrs vs. >38 yrs); Difference in Live Birth Rates = -2.3, 95% CI 2-sided [-6.5 to 1.9]

4. Secondary Outcome: Number of Participants With Moderate or Severe Ovarian Hyperstimulation Syndrome (OHSS)
Description: Grade II (moderate OHSS) is characterized by distinct ovarian cysts (ovary size 8-10 cm), accompanied by abdominal pain and tension, nausea, vomiting, diarrhea.
  Grade III (severe OHSS) is characterized by enlarged cystic ovaries (ovary size >10 cm), accompanied by ascites and occasionally hydrothorax. Abdominal tension and pain may be severe. Pronounced hydrothorax together with an abdominal cavity filled with cysts and fluid elevating the diaphragm, may cause severe breathing difficulties. Large quantities of fluid inside the cysts and in the peritoneal and pleural cavities cause hemoconcentration and increased blood viscosity. In rare cases, the syndrome may further be complicated by the occurrence of thromboembolic phenomena.
Time Frame: Up to approximately 1 month after oocyte pick-up
Population: All-Subjects-Treated (AST) Group, defined as all participants who received 1 or more dose(s) of SCH 900962 or recFSH. Participants were grouped according to the active treatment they actually received.
Measure: Number; unit: participants
Arm/Group | Single Injection of 150 µg SCH 900962/MK-8962 | Daily 300 IU recFSH
Number analyzed (Participants) | 692 | 698
participants | 5 | 10
Statistical Analysis 1: Comparison: Single Injection of 150 µg SCH 900962/MK-8962 vs Daily 300 IU recFSH; Test type: Superiority or Other; p = 0.30, Fisher Exact

5. Secondary Outcome: Number of Participants Who Cancelled the Cycle Due to a (Serious) Adverse Event
Description: The number of participants who started stimulation but did not undergo embryo transfer due to (S)AEs will be compared between the treatment groups.
Time Frame: Up to time of embryo transfer (maximum of 24 days after start of study drug)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Single Injection of 150 µg SCH 900962/MK-8962 | Daily 300 IU recFSH
Number analyzed (Participants) | 692 | 698
participants | 5 | 6
Statistical Analysis 1: Comparison: Single Injection of 150 µg SCH 900962/MK-8962 vs Daily 300 IU recFSH; Test type: Superiority or Other; p > 0.999, Fisher Exact

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were reported for both pretreatment and active treatment periods of the Intervention Phase of the study, inclusive. AEs for the Follow-up Period include events reported by the mother/fetus/infant (up to 4-12 weeks after birth).
Description: Safety Population: All Subjects Treated, defined as all participants who received 1 or more dose(s) of SCH 900962 or recFSH. Participants were grouped according to the active treatment they actually received. Three participants randomized to SCH900962 were treated with recFSH, and 1 participant randomized to recFSH was treated with SCH900962.
Groups:
- Single Injection of 150 µg SCH 900962/MK-8962-Follow-up: Participants who received a single injection of 150 ug SCH 900962 (MK-8962) on Stimulation Day 1 and 7 injections with placebo-recFSH from Stimulation Days 1-7 during Intervention Period and became pregnant.
- Daily 300 IU recFSH -Follow-up: Participants who received a single injection of placebo SCH 900962 (MK-8962) on Stimulation Day 1 and 7 injections of recFSH from Stimulation Days 1-7 during Intervention Period and became pregnant.
Arm/Group | Single Injection of 150 µg SCH 900962/MK-8962 | Daily 300 IU recFSH | Single Injection of 150 µg SCH 900962/MK-8962-Follow-up | Daily 300 IU recFSH -Follow-up
Serious Adverse Events (participants affected / at risk) | 4/692 | 19/698 | 110/154 | 112/167
Other Adverse Events (participants affected / at risk) | 267/692 | 262/698 | 94/154 | 105/167
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Injection of 150 µg SCH 900962/MK-8962 (N=692) | Daily 300 IU recFSH (N=698) | Single Injection of 150 µg SCH 900962/MK-8962-Follow-up (N=154) | Daily 300 IU recFSH -Follow-up (N=167)
CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABORTION INFECTED (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
FOREIGN BODY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OVERDOSE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CEREBRAL ISCHAEMIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEMIANOPIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ABORTION MISSED (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
ECTOPIC PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 8 (8) | 0 (0) | 0 (0)
OVARIAN HYPERSTIMULATION SYNDROME (Reproductive system and breast disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0)
INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THROMBOCYTOPENIA NEONATAL (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRADYCARDIA NEONATAL (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FOETAL HEART RATE DECELERATION (Cardiac disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
VENTRICULAR HYPERTROPHY (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACCESSORY AURICLE (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANKYLOGLOSSIA CONGENITAL (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 6 (6)
ARNOLD-CHIARI MALFORMATION (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATRIAL SEPTAL DEFECT (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
BRAIN MALFORMATION (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHORDEE (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CONGENITAL AORTIC ANOMALY (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONGENITAL CARDIOVASCULAR ANOMALY (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
CONGENITAL CENTRAL NERVOUS SYSTEM ANOMALY (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONGENITAL CHOROID PLEXUS CYST (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
CONGENITAL CYSTIC DISEASE OF LIVER (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONGENITAL GENITAL MALFORMATION MALE (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CONGENITAL HYDRONEPHROSIS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
CONGENITAL HYPOTHYROIDISM (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONGENITAL INGUINAL HERNIA (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONGENITAL MELANOCYTIC NAEVUS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONGENITAL ORAL MALFORMATION (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
CONGENITAL PIGMENTATION DISORDER (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
CONGENITAL PYELOCALIECTASIS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
CONGENITAL TORTICOLLIS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DACRYOSTENOSIS CONGENITAL (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (5)
DEAFNESS CONGENITAL (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DERMOID CYST (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSMORPHISM (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
EXOMPHALOS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 5 (5) | 3 (4)
FALLOT'S TETRALOGY (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FOETAL CYSTIC HYGROMA (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HAEMANGIOMA CONGENITAL (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 4 (4) | 6 (6)
HIGH ARCHED PALATE (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HIP DYSPLASIA (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 6 (7)
HOODED PREPUCE (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYDROCELE (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOPLASTIC LEFT HEART SYNDROME (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOSPADIAS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INTESTINAL MALROTATION (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LARYNGOMALACIA (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PATENT DUCTUS ARTERIOSUS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 4 (4) | 1 (2)
PECTUS EXCAVATUM (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PHIMOSIS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLAGIOCEPHALY (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
PULMONARY ARTERY STENOSIS CONGENITAL (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RESPIRATORY TRACT MALFORMATION (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEPTUM PELLUCIDUM AGENESIS (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKULL MALFORMATION (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SPINA BIFIDA (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TALIPES (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
TELANGIECTASIA CONGENITAL (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TRISOMY 13 (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TRISOMY 18 (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
TRISOMY 21 (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
TRISOMY 22 (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URACHAL ABNORMALITY (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VENTRICULAR SEPTAL DEFECT (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FUNCTIONAL GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TEMPERATURE REGULATION DISORDER (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERBILIRUBINAEMIA NEONATAL (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
APPENDICITIS PERFORATED (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CHORIOAMNIONITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENDOMETRITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HERPES VIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
KIDNEY INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PARONYCHIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEPSIS NEONATAL (Infections and infestations) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
FOETAL HEART RATE ABNORMAL (Investigations) | 0 (0) | 0 (0) | 6 (6) | 5 (5)
FOETAL HEART RATE DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FOETAL NON-STRESS TEST ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FEEDING DISORDER NEONATAL (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3) | 2 (2)
HYPOGLYCAEMIA NEONATAL (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RETROGNATHIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CEREBRAL VENTRICLE DILATATION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTRAVENTRICULAR HAEMORRHAGE NEONATAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MIGRAINE WITH AURA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ARRESTED LABOUR (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 16 (16) | 13 (13)
BREECH PRESENTATION (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 12 (12) | 14 (14)
CEPHALO-PELVIC DISPROPORTION (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
CERVICAL INCOMPETENCE (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DISCORDANT TWIN (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FAILED INDUCTION OF LABOUR (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
FOETAL DEATH (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FOETAL DISTRESS SYNDROME (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
FOETAL GROWTH RESTRICTION (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
FOETAL MACROSOMIA (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 3 (3)
FOETAL MALPRESENTATION (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GESTATIONAL DIABETES (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
GESTATIONAL HYPERTENSION (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
HAEMORRHAGE IN PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
HELLP SYNDROME (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
JAUNDICE NEONATAL (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 4 (5) | 1 (1)
LOW BIRTH WEIGHT BABY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
MECONIUM IN AMNIOTIC FLUID (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MULTIPLE PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OLIGOHYDRAMNIOS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
PERIPARTUM CARDIOMYOPATHY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PLACENTA PRAEVIA (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (3) | 5 (5)
PLACENTA PRAEVIA HAEMORRHAGE (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
POSTPARTUM HAEMORRHAGE (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PRE-ECLAMPSIA (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 7 (7) | 7 (7)
PREGNANCY WITH ADVANCED MATERNAL AGE (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PREMATURE BABY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 15 (25) | 17 (28)
PREMATURE LABOUR (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (3) | 8 (8)
PREMATURE RUPTURE OF MEMBRANES (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 4 (4) | 6 (6)
PREMATURE SEPARATION OF PLACENTA (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
PREVIOUS CAESAREAN SECTION (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 11 (11) | 14 (14)
PROLONGED LABOUR (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROLONGED PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
RETAINED PLACENTA OR MEMBRANES (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
SMALL FOR DATES BABY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
STILLBIRTH (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THREATENED LABOUR (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
TRANSVERSE PRESENTATION (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
TWIN PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 10 (10) | 11 (11)
UMBILICAL CORD AROUND NECK (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UTERINE CERVICAL LACERATION DURING LABOUR (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VASA PRAEVIA (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WEIGHT DECREASE NEONATAL (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
BLADDER DYSFUNCTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CERVIX DISORDER (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CERVIX OEDEMA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PELVIC PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SHORTENED CERVIX (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATELECTASIS NEONATAL (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHOPULMONARY DYSPLASIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
IMMATURE RESPIRATORY SYSTEM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFANTILE APNOEIC ATTACK (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEONATAL ASPIRATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEONATAL RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 7 (8) | 6 (8)
NEONATAL RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
PULMONARY OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TRANSIENT TACHYPNOEA OF THE NEWBORN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABORTION INDUCED (Surgical and medical procedures) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
CAESAREAN SECTION (Surgical and medical procedures) | 0 (0) | 0 (0) | 8 (8) | 5 (5)
MYOMECTOMY (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
SELECTIVE ABORTION (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Injection of 150 µg SCH 900962/MK-8962 (N=692) | Daily 300 IU recFSH (N=698) | Single Injection of 150 µg SCH 900962/MK-8962-Follow-up (N=154) | Daily 300 IU recFSH -Follow-up (N=167)
NAUSEA (Gastrointestinal disorders) | 47 (50) | 33 (36) | 10 (10) | 15 (15)
POST PROCEDURAL COMPLICATION (Injury, poisoning and procedural complications) | 61 (64) | 69 (72) | 5 (7) | 4 (4)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 98 (101) | 83 (86) | 13 (15) | 18 (20)
HEADACHE (Nervous system disorders) | 73 (98) | 73 (101) | 6 (10) | 11 (11)
ABORTION MISSED (Pregnancy, puerperium and perinatal conditions) | 29 (29) | 39 (39) | 0 (0) | 0 (0)
PELVIC DISCOMFORT (Reproductive system and breast disorders) | 52 (57) | 57 (66) | 4 (5) | 6 (6)
CONSTIPATION (Gastrointestinal disorders) | 21 (23) | 22 (22) | 17 (19) | 20 (24)
DYSPEPSIA (Gastrointestinal disorders) | 4 (4) | 14 (15) | 9 (13) | 17 (17)
FLATULENCE (Gastrointestinal disorders) | 4 (4) | 2 (2) | 9 (11) | 8 (8)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 (2) | 1 (1) | 16 (17) | 15 (18)
URINARY TRACT INFECTION (Infections and infestations) | 14 (14) | 7 (7) | 9 (9) | 5 (5)
PERINEAL LACERATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 8 (8) | 14 (14)
AFTERBIRTH PAIN (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 11 (13) | 11 (12)
GESTATIONAL DIABETES (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 15 (16) | 14 (14)
JAUNDICE NEONATAL (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 31 (33) | 27 (30)
PREMATURE BABY (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 14 (20) | 10 (13)
VOMITING IN PREGNANCY (Pregnancy, puerperium and perinatal conditions) | 25 (28) | 31 (35) | 10 (11) | 9 (9)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 9 (9) | 8 (8)
NEONATAL RESPIRATORY DISTRESS SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 8 (9) | 4 (5)
ANAEMIA (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 7 (7) | 14 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agreed not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agreed to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report(s) any results of the trial.